CLINICAL TRIAL: NCT06493786
Title: Identification of Olfactory Biomarkers of Skin Cancer From Skin Odor Samples: a Pilot Study
Acronym: SCENT-SKIN-001
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Collaborators: SenseBioTek Health-Care (Unknown); ESPCI Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A00450-47
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Identify Volatile Biomarkers Specific to Malignant Melanoma, Basal Cell Carcinoma and Squamous Cell Carcinoma; Verify That the Volatile Biomarkers Identified Derive From Metabolic Changes in Body Odour and Not Just From Changes in the Surface of Cancerous Lesions
Keywords: collection of body odor samples; volatile biomarkers; various skin cancers
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Malignant melanoma (MM) (Other): For each group of patients (MM, CBC*, CE), the chromatographic profiles of cutaneous VOCs (nature of molecules and content) will be described and compared as follows:
  healthy areas (excluding contralateral areas) versus healthy areas of matched healthy subjects, by area and overall.
  * For the BCC group, the same analyses will be performed for the 3 BCC categories: superficial BCC, nodular BCC, infiltrating BCC.
  Interventions: Other: Collection of body odor samples
- Basocellular carcinoma (BCC) (Other): For each group of patients (MM, CBC*, CE), the chromatographic profiles of cutaneous VOCs (nature of molecules and content) will be described and compared as follows:
  healthy areas (excluding contralateral areas) versus healthy areas of matched healthy subjects, by area and overall.
  * For the BCC group, the same analyses will be performed for the 3 BCC categories: superficial BCC, nodular BCC, infiltrating BCC.
  Interventions: Other: Collection of body odor samples
- Epidermoid carcinoma (EC) (Other): For each group of patients (MM, CBC*, CE), the chromatographic profiles of cutaneous VOCs (nature of molecules and content) will be described and compared as follows:
  healthy areas (excluding contralateral areas) versus healthy areas of matched healthy subjects, by area and overall.
  * For the BCC group, the same analyses will be performed for the 3 BCC categories: superficial BCC, nodular BCC, infiltrating BCC.
  Interventions: Other: Collection of body odor samples
- Healthy volunteers (Other): For each group of patients (MM, CBC*, CE), the chromatographic profiles of cutaneous VOCs (nature of molecules and content) will be described and compared as follows:
  healthy areas (excluding contralateral areas) versus healthy areas of matched healthy subjects, by area and overall.
  * For the BCC group, the same analyses will be performed for the 3 BCC categories: superficial BCC, nodular BCC, infiltrating BCC.
  Interventions: Other: Collection of body odor samples

INTERVENTIONS:
Other: Collection of body odor samples — Skin odor is collected using polymer sticks, placed in contact with the skin for approximately 1 hour.
  In this study, odor collection will be carried out on the thigh, forearm, armpit, neck and, if applicable, on the cancerous lesion.

SUMMARY:
The aim of this research is to determine which volatile organic compounds (odors) are associated with different skin cancers.

To this end, odor samples will be taken from various parts of the body, from patients with skin cancers and from "healthy" subjects who have no skin cancer.

The various samples collected will be analyzed in the laboratory, and compared with each other, to determine whether there is a specific "smell" for the main types of skin cancer.

DETAILED DESCRIPTION:
The SCENT-SKIN-001 exploratory study aims to identify olfactory biomarkers associated with skin cancers. Body odor samples will be collected from patients with skin cancers at the level of the skin lesion, the area contralateral to the skin lesion, the axillary fossa, the neck, the forearm and the inner thigh, and from healthy subjects at the level of the axillary fossa, the neck, the forearm and the inner thigh. Samples will be analyzed by thermodesorption followed by fully two-dimensional gas chromatography coupled to time-of-flight mass spectrometry (TD-GCxGC/ToFMS). This sample characterization method can separate a much higher number of compounds than the simple GC-MS technique. It has been developed in collaboration with the team at the Laboratoire de Sciences Analytiques, Bioanalytiques et Miniaturisation (LSABM), École Supérieure de Physique et de Chimie Industrielle de la Ville de Paris (ESPCI Paris), and is the subject of a doctoral thesis in analytical chemistry. As part of this analytical method, we have developed a skin VOC sampling device. This is designed to avoid any form of contamination by environmental factors that could influence sample quality.

The study will be carried out on patients newly diagnosed with malignant melanoma, basal cell carcinoma or squamous cell carcinoma, and on "healthy" subjects with no skin cancer.

60 skin cancer patients (20 with Malignant Melanoma, 20 with Basal Cell Carcinoma and 20 with Epidermoid Carcinoma) and 20 to 60 healthy subjects will be included in the study. Thus, the study will involve 80 to 120 people.

The study will be carried out in French hospitals, as well as in a center authorized by the Agence Régionale de Santé (ARS) to conduct clinical trials on healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* For patients

  1. Adult patient (age ≥ 18 years),
  2. Patient with a diagnosis of skin cancer of the malignant melanoma, basal cell carcinoma or squamous cell carcinoma type, established by in vivo imaging of the confocal microscopy or LC-OCT type, more than 24 hours old (definitive confirmation being made by anatomopathological examination of the postoperative excision specimen),
  3. Patient with a lesion located on a flat surface measuring at least 3 cm by 2 cm,
  4. Patient who has not applied any cosmetic products, such as deodorant, perfume, perfumed cream or soap, or hair care products, in the 24 hours prior to sampling,
  5. Patient who has not handled odorous substances (e.g. household products, paints) in the 24 hours prior to sampling,
  6. Patient who has not eaten a meal (or flavored substances such as drinks or sweets) within 2 hours of sampling,
  7. Patient able to read, understand and give documented informed consent,
  8. Patient willing and able to comply with protocol requirements for the duration of the study,
  9. Patient affiliated or entitled to a social security scheme,
  10. for patients of childbearing potential, negative pregnancy test at inclusion.
* For healthy subjects

  1. Adult subject (age ≥ 18 years),
  2. Subject who, in the judgement of the dermatological investigator, does not have a suspicious or pre-cancerous skin lesion suggestive of skin cancer.
  3. Subject who has not applied any cosmetic products, such as deodorant, perfume, perfumed cream or soap, or hair care products, in the 24 hours prior to sampling,
  4. Subject not to have handled odorous substances (e.g. household products, paints) in the 24 hours prior to sampling,
  5. Subject not having eaten a meal (or flavored substances such as drinks or sweets) in the 2 hours prior to sampling,
  6. Subject able to read, understand and give documented informed consent,
  7. Willing and able to comply with protocol requirements for the duration of the study.
  8. Subject affiliated or entitled to a social security plan,
  9. For subjects of childbearing potential, negative pregnancy test at inclusion.

Exclusion Criteria:

1. Patient or subject who has expressed opposition to participation in the study,
2. Patient or subject under guardianship, deprived of liberty, under psychiatric care or hospitalized in a health or social institution,
3. Patient or subject linguistically unable to understand the terms of the study,
4. Pregnant and/or breast-feeding and/or likely to become pregnant,
5. Patient or subject with a known allergy to adhesive dressings,
6. Patient or subject with inflammatory skin disease, infectious skin disease or any other suspicious or pre-cancerous skin lesion,
7. Patient or subject with a known history of progressive cancer within the last five (5) years,
8. Patient or subject with an additional condition which, in the opinion of the investigator, may interfere with the evaluation of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of chromatographic profiles of skin VOCs | 12 months
  For each group of patients (MM, CBC*, CE), the chromatographic profiles of cutaneous VOCs (nature of molecules and content) will be described and compared as follows:
  healthy areas (excluding contralateral areas) versus healthy areas of matched healthy subjects, by area and overall.
  * For the BCC group, the same analyses will be performed for the 3 BCC categories: superficial BCC, nodular BCC, infiltrating BCC.

IPD SHARING:
Plan to Share IPD: No